CLINICAL TRIAL: NCT05926856
Title: Comparison of the Fluorescent Visualization of the Extrahepatic Biliary Tract Between Two Injection Protocols
Brief Title: High Quality Fluorescent Cholangiography
Acronym: HQFC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Chihua Fang,MD, Professor, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20230420
Record Dates: First submitted 2023-06-02; First posted 2023-07-03 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Extrahepatic Biliary Tree Injury
Keywords: icg; fluorescent cholangiograph
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 day before surgery (Active Comparator): 0.25mg/kg Indocyanine Green will be administered 1 day before surgery
  Interventions: Drug: Indocyanine green
- 45 min before surgery (Experimental): 0.05mg Indocyanine Green will be administered 45minutes before surgery
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — Indocyanine Green 25mg kit for injection

SUMMARY:
The goal of this randomized controlled trial is to compare the quality of extrahepatic biliary fluorescent visualization under two injection protocols to optimize extrahepatic biliary cholangiography.

DETAILED DESCRIPTION:
Biliary fluorescence imaging is widely used to identify the extrahepatic biliary tract during laparoscopic cholecystectomy. However, fluorescent developer Indocyanine Green（ICG） still lacks standardization, and not every visualization of the extrahepatic biliary tract is satisfactory. Some research groups have shown that injection of ICG 1 day before surgery can achieve the best fluorescence imaging of the biliary tract, but some research groups have suggested that injection of a very low dose of ICG 45 minutes before surgery can improve the satisfaction of fluorescence imaging. However, no study compares the quality of biliary fluorescence imaging between the two injection protocols. This study will compare the fluorescence imaging effects of the two schemes to obtain the best injection scheme at present and standardize the use of icg.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has indications for cholecystectomy and requires laparoscopic treatment；
2. No biliary obstruction or cholestasis was found during preoperative examination；3.Volunteer to participate in this clinical trial and sign written informed consent.

Exclusion Criteria:

1. Patients who require emergency surgical treatment；
2. Patients with malignant tumors of the biliary tract；
3. Patients with a history of abdominal surgery；
4. Patients who are allergic to indocyanine green or iodine contrast agents；5.Patients participating in one or more other clinical trials simultaneously；

6.Patients who have received medication that affects bile excretion within 2 weeks before surgery； 7.Other situations that have been judged unsuitable for inclusion by researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Common bile duct-to-liver fluorescence intensity ratio | Intraoperative (The beginning of the surgery)
  Common bile duct-to-liver fluorescence intensity ratio

CONTACTS AND LOCATIONS:
Overall Officials: Jian Yang, MD, Principal Investigator — Zhujiang Hospital
Locations (1):
- Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No